CLINICAL TRIAL: NCT03163901
Title: The Effect of OMT on Functional Outcomes and Anti-inflammatory Biomarkers in Mild to Moderate Traumatic Brain Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Michigan State University (Other)
Collaborators: American Osteopathic Association (Other)
Responsible Party: Principal Investigator, Rebecca Wyatt, Assistant Professor, Michigan State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: i053814
Record Dates: First submitted 2017-05-15; First posted 2017-05-23 (Actual); Last update posted 2020-06-24 (Actual); Status verified 2020-06

CONDITIONS: Vestibular Disorder; Headache; Traumatic Brain Injury
Keywords: traumatic brain injury
MeSH Terms: conditions — Vestibular Diseases; Headache; Brain Injuries, Traumatic | interventions — Manipulation, Osteopathic

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Treatment groups (Active Comparator): To recruit and organize patients with TBI enrolled in a standard rehabilitation program into three groups ((a) treatment group receiving OMT; (b) control group A receiving sham treatment; and (c) control group B receiving neither OMT nor sham treatment) in order to assess the feasibility and adherence to the protocol and determine participation and attrition rates in preparation for a larger study.
  Interventions: Other: Osteopathic Manipulative Treatment
- Effect of OMT on clinical outcome measures (Other): Clinical outcome measures including Neurocom Balance Manager assessments (Modified Clinical Test of Sensory Interaction and Balance; Stability Evaluation Test; Rhythmic Weight Shift; Limits of Stability), Vestibular Oculomotor Screen, Motion Sensitivity Test, as well as questionnaires such as the Headache Impact Test (HIT-6), Dizziness Handicap Inventory, and the more general quality of life measures (dressing; bathing; medication management, etc. as assessed by the SF 36 QOL questionnaire).
  Interventions: Other: Osteopathic Manipulative Treatment
- Anti-inflammatory Biomarkers (No Intervention): to analyze urine and plasma samples collected from the three groups of participants: urine and plasma samples one hour before, plasma samples one hour after and 48 hours after treatment for alterations in the levels of low molecular weight compounds or protein components to identify potential biomarkers that may correlate with the TBI condition and/or the OMT.
- Infrastructure development (No Intervention): to establish the infrastructure for the recording, management, and extraction of clinical data and to estimate effect sizes and variability in key outcome measures so that a larger, longer term study can be planned with sufficient statistical power to identify significant results.

INTERVENTIONS:
Other: Osteopathic Manipulative Treatment — OMT techniques applied in the thoracic spine soft tissue, cervical spine soft tissue, suboccipital release, occipital condyle condylar decompression, and cranial venous sinus release.
  Other Names: OMT
  Arms: Effect of OMT on clinical outcome measures; Treatment groups

SUMMARY:
Test the hypothesis that a certain set of osteopathic manipulation procedures preformed on patients with mild to moderate traumatic brain injury will result in accelerated rates of recovery assessed using vestibular function tests, quality of life questionnaires and measurements of the levels of anti-inflammatory metabolite and protein biomarkers in the blood and urine.

DETAILED DESCRIPTION:
This project proposes to test the hypothesis that a certain set of osteopathic manipulative treatment (OMT) procedures performed on patients with mild to moderate traumatic brain injury (TBI) will result in accelerated rates of recovery as assessed using vestibular function tests, patient response on quality of life questionnaires, and measurements of the levels of anti-inflammatory metabolite and protein biomarkers in urine and blood. The OMT techniques, performed ensemble (as a set) and in sequence, will encompass: (a) soft tissue to the upper-mid thoracic spine; (b) soft tissue to the cervical spine; (c) suboccipital release; (d) condylar decompression; and (e) cranial venous sinus release. The key clinical outcome measures will include Neurocom Balance Manager assessments (Modified Clinical Test of Sensory Interaction and Balance; Stability Evaluation Test; Rhythmic Weight Shift; Limits of Stability), Vestibular Oculomotor Screen, Motion Sensitivity Test, as well as questionnaires such as Headache Impact Test (HIT-6), Dizziness Handicap Inventory, and the more general quality of life measures (dressing, bathing, medication management, etc. as assessed by the SF 36 QOL questionnaire).

A unique and trail blazing aspect of our proposed work is to screen for biochemical alterations in the plasma and urine of these patients following administration of OMT and to correlate these changes with vestibular function tests and other clinical parameters that may shed light on the biological mechanism(s) underlying the OMT. The impact of our proposed research lies in our attempt to establish a foundation for the basis of using OMT procedures to accelerate recovery of patients following mild to moderate brain injury and to find correlations between cognitive functions, biochemical markers, and self-reported assessments of quality of life.

The successful achievement of positive outcomes in this project will serve as the basis for our future efforts to seek funding from the National Institutes of Health for recruitment of larger numbers of subjects in a multi-center research effort.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of mild to moderate traumatic brain injury
* Chief complaint of headache and/or dizziness
* 18 years or older
* Medically stable/free from acute infection or fever
* Not a danger to self or others
* Not actively engaged in substance abuse
* Minimum Ranchos Los Amigos Level of 4 (http://www.traumaticbraininjury.com/symptoms-of-tbi/).

Exclusion Criteria:

* Minors below age of 18
* Any acute fracture or bleeding
* Head, neck or back wounds that would prevent OMT treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2017-09-18 (Actual); Primary Completion 2020-02-29 (Actual); Study Completion 2020-02-29 (Actual)

PRIMARY OUTCOMES:
Change from baseline Neurocom Balance Manager assessment in 12 weeks after OMT | 12 weeks
  Participants will be evaluated prior to treatment on the Neurocom Balance Manager. Reassessment done at 12 week. The balance score will be recorded.
Change of baseline Headache Impact Test (HIT-6) scores after 12 weeks of OMT | 12 weeks
  Participants will be given the HIT-6 questionnaire at 0 and12 weeks. The scores will be recorded.

SECONDARY OUTCOMES:
Change in Anti-inflammatory Biomarker after 12 weeks of OMT or sham treatment | 12 weeks
  Urine sample will be taken one hour prior to initial OMT or sham treatment and again at12 weeks. Plasma samples will be taken one hour prior to OMT/sham treatment and 48 hours after treatment this will be done at week 0, 6 and 12. The anti-inflammatory biomarkers will be recorded and compared (before/after treatment) to see if they levels decrease after OMT treatments

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Wyatt, DO, Principal Investigator — Assistant Professor at Michigan State University
Locations (1):
- Origami Brain Injury Rehabilitation Center, Mason, Michigan, United States